CLINICAL TRIAL: NCT06301282
Title: Electroencephalographic Signatures of Neuropsychiatric Fluctuations in Parkinson's Disease and the Temporal Dynamics of Their Dopaminergic Modulation
Brief Title: Electroencephalographic Signatures of Neuropsychiatric Fluctuations in Parkinson's Disease
Acronym: Transition
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Vanessa Fleury, Principal Investigator, University Hospital, Geneva
Other Study IDs: 2021-02341
Record Dates: First submitted 2024-01-16; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: assessment during the transition between OFF-levodopa (i.e. withdrawal of levodopa phase) and ON-levodopa (i.e. effect of Levodopa phase)states — Electroencephalographic measurements are taken during both motor and non-motor assessments while the transition between the OFF-levodopa and ON-levodopa states occurs

SUMMARY:
Dopaminergic replacement therapy while efficient at reducing symptoms of Parkinson's disease is however often associated with motor and non-motor fluctuations which have a severe impact on patient quality of life. To date, the interplay between cortical activity linked to motor and non-motor symptoms and Parkinson's disease fluctuations linked to dopaminergic medication remain poorly understood.

The aim of the study is to characterize the cortical electroencephalographic oscillatory correlates of Parkinson's disease motor and non-motor fluctuations and the temporal dynamics of their dopaminergic modulation.

For this purpose, the investigators will apply an innovative approach using the differential non-linear temporal dynamics of motor and non-motor state during the transition from the dopaminergic withdrawal phase (i.e. OFF-levodopa state) to the dopaminergic effect phase (i.e. ON-levodopa state) following an acute levodopa administration.

This research will allow to precisely disentangle the network dynamics subtending motor and non-motor symptoms of Parkinson's disease as well as precisely identify the electroencephalographic spectral modulations explaining the neuropsychiatric effects of levodopa. The identification of such biomarkers could pave the way toward innovative therapeutic approaches such as neurofeedback and transmagnetic stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease (PD) based on United Kingdom PD Society Brain Bank Criteria
* Patients in the PD phase called "fluctuation stage". PD can be defined according to the four following disease stages: de novo stage (i.e. at the time of diagnosis, dopamine replacement therapy not yet introduced), honeymoon stage (i.e. dopamine replacement therapy compensates PD symptoms), motor and non-motor fluctuations stage (fluctuations in the clinical effect of the dopamine replacement therapy) and the decline phase (i.e. onset of cognitive impairment and falls).
* Presence of motor and non-motor fluctuations are based on:

  * For motor fluctuations: a score of 1 on item 4.1 and/or 1 on item 4.3 of the Movement Disorder Society Unified Parkinson's Disease Rating Scale IV
  * For non-motor fluctuations: a score of 2 on item III of the Behavioral Assessment of PD
* To be on dopaminergic replacement therapy. The daily dose of dopaminergic replacement therapy will be converted into a common unit (levodopa equivalent daily dose) to get an idea of the dopaminergic replacement therapy dose needed per day for each patient

The course of PD, and in particular the time of each PD phase, is very variable from one patient to another. A precise duration of illness can therefore not be included in the inclusion criteria. The dose of dopaminergic replacement therapy required for each patient is also extremely variable from one patient to another and cannot be included in the inclusion criteria.

Healthy controls will be subjects:

• Without any known central nervous system (CNS) lesion or CNS clinical signs on examination

Exclusion Criteria:

* Age greater than 80 years
* Dementia or mild cognitive impairment based on a score <24 on the MOntreal Cognitive Assessment,
* Ongoing depression with suicidal ideation,
* Any clinically meaningful non-stable renal, hepatic, cardiovascular, respiratory, cerebrovascular disease or other serious progressive physical diseases,
* Participating in a pharmacological study,
* Intolerable "OFF-levodopa" states when the effects of the PD medication wear off (e.g., severe pain, anxiety, depression at the end of the dose or in the morning upon waking),
* Inability to provide informed consent (legal guardianship),
* Inability to speak or read French.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's Disease (PD) patients will be recruited from the outpatient movement disorder clinic of the Neurology Department at the Geneva University Hospital (HUG). Patients, who participated in previous studies and who are now followed-up by private physicians, could also be contacted by trained members of the clinic/research staff to propose the study.
  Flyers with a brief explanation of the project could also be distributed to the physicians for inviting patients to consider participating and reach out to a staff member for further information.
  Healthy controls will be recruited among the spouse of patients and through advertisement placed in the HUG and the University Medical Centre.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of electroencephalographic resting-state oscillatory activity with neuropsychiatric clinical scores during the levodopa challenge | 90 minutes
  Correlation between electroencephalographic data (frequency, time, cortical location) and neuropsychiatric scores (neuropsychiatric fluctuation score, anxiety and depression scores, apathy score, bradyphrenia score)

SECONDARY OUTCOMES:
Correlation of electroencephalographic resting-state oscillatory activity with motor scores during the levodopa challenge | 90 minutes
  Correlation of electroencephalographic resting-state oscillatory activity with motor scores (akinesia, rigidity)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Fleury, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital, Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No